CLINICAL TRIAL: NCT06920875
Title: The Effect of 10-Week Imagery and Breathing Exercises on 200-Meter Swimming Performance, Mental Toughness, and Heart-Mind Coherence in Swimmers: A Randomized Controlled Trial
Brief Title: Effects of Imagery and Breathing Exercises on Swimmers' Performance, Mental Toughness, and Heart-Mind Coherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-60116787-020-666811
Record Dates: First submitted 2025-03-16; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Athletic Performance; Mental Toughness; Coherence (Heart-Mind Synchronization)
Keywords: Swimming; Imagery; Mental Toughness; Coherence; Heart Rate Variability; Breathing Exercises; Sports Psychology; Athletic Performance; Mental Training
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, parallel-group, pre-test post-test design.
Masking Description: None (Open Label) (The manuscript does not mention blinding; assumed as open-label since participants and researchers likely knew the group assignments due to the nature of the intervention.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imagery and Breathing Exercises (Experimental): Participants received a 10-week intervention of imagery and breathing exercises in addition to standard physical training.
  Interventions: Behavioral: Imagery and Breathing Exercises
- Standard of care (No Intervention): Participants received only standard physical training without additional mental training.

INTERVENTIONS:
Behavioral: Imagery and Breathing Exercises — Participants performed daily imagery and breathing exercises before bedtime for 10 weeks. The protocol involved a 4-second inhale through the nose and a 4-second exhale through the mouth while visualizing a 200-meter freestyle swim with detailed attention to technique and performance. A 6-day training period was provided to teach the techniques, and participants received daily reminders and feedback via a WhatsApp group.
  Arms: Imagery and Breathing Exercises

SUMMARY:
This randomized controlled trial aimed to investigate the effects of a 10-week imagery and breathing exercise intervention on 200-meter freestyle swimming performance, mental toughness, and heart-mind coherence in swimmers. Nineteen licensed swimmers aged 13-18 years were randomly assigned to an experimental group (n=9) receiving imagery and breathing exercises or a control group (n=10) receiving only standard physical training. Outcomes were measured using the 200-meter freestyle swimming time, the Sports Mental Toughness Questionnaire (SMTQ), and heart-mind coherence via the Inner Balance HeartMath device. The intervention significantly improved mental toughness and swimming performance in the experimental group compared to the control group, with a trend toward improved heart-mind coherence.

DETAILED DESCRIPTION:
The study was conducted at the facilities of Pamukkale Üniversitesi Mensupları Spor Kulübü Yüzme Takımı in Denizli, Türkiye. Participants underwent a pre-test/post-test design with the following measures: 200-meter freestyle swimming performance, mental toughness (assessed via the Sports Mental Toughness Questionnaire), and heart-mind coherence (measured using the Inner Balance HeartMath device for real-time biofeedback of heart rate variability [HRV]). The experimental group participated in a 10-week intervention involving daily imagery and breathing exercises performed before bedtime, following a structured protocol (4-second inhale through the nose, 4-second exhale through the mouth, while imagining a 200-meter swim with detailed visualization). The intervention included a 6-day training period on techniques, followed by 10 weeks of daily practice, with reminders and feedback provided via a WhatsApp group. The control group continued standard physical training without additional mental training. Data were analyzed using a two-way repeated measures ANOVA, with post-hoc Bonferroni tests, and a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-18 years.
* Licensed and actively engaged in competitive swimming.
* No serious injuries in the past 6 months.
* Parental consent obtained for participants under 18 years.

Exclusion Criteria:

* Diagnosis of heart disease or respiratory system disorders.
* Psychiatric diagnosis or ongoing psychological treatment.
* Serious injury or surgery within the past 6 months.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
200-Meter Freestyle Swimming Performance | Baseline (pre-test) and 10 weeks (post-test).
  time to complete a 200-meter freestyle swim, measured in seconds.
Mental Toughness | Baseline (pre-test) and 10 weeks (post-test).
  Assessed using the Sports Mental Toughness Questionnaire (SMTQ), with scores indicating levels of mental toughness. The Sports Mental Toughness Questionnaire (SMTQ) is a 14-item scale measuring mental toughness across the subdomains of confidence, constancy, and control, with scores ranging from 14 to 56. Higher scores indicate greater mental toughness, reflecting a more positive psychological profile in athletes.
Heart-Mind Coherence | Baseline (pre-test) and 10 weeks (post-test).
  Measured using the Inner Balance HeartMath device to assess heart rate variability (HRV)

SECONDARY OUTCOMES:
Maximum Coherence Values | Baseline (pre-test) and 10 weeks (post-test).
  Maximum coherence levels achieved during measurement sessions, assessed via the Inner Balance HeartMath device.
Balance Performance | Baseline (pre-test) and 10 weeks (post-test).
  Assessed as part of the study hypothesis, though specific measurement tools are not detailed in the manuscript.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No